CLINICAL TRIAL: NCT06450613
Title: Cost-effectiveness of Radiofrequency Ablation vs. Percutaneous Ethanol Injection for Early-stage HCC in a Resource-poor Setting - a Randomized Trial
Brief Title: Cost-effectiveness of RFA vs. PEI for Early-stage HCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 68277917.4.0000.0071
Record Dates: First submitted 2023-11-23; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2021-03

CONDITIONS: Cost Effectiveness; Exposure to Radiofrequency
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- percutaneous ethanol injection (Other): early-stage hepatocellular carcinoma within the Milan criteria, listed for LT and with indication for neoadjuvant treatment were eligible for enrollment submitted to percutaneous ethanol injection
  Interventions: Other: percutaneous ethanol injection
- Radiofrequency ablation (Other): early-stage hepatocellular carcinoma within the Milan criteria, listed for LT and with indication for neoadjuvant treatment were eligible for enrollment submitted to Radiofrequency ablation
  Interventions: Device: radiofrequency ablation

INTERVENTIONS:
Device: radiofrequency ablation — HCC Radiofrequency ablation
  Arms: Radiofrequency ablation
Other: percutaneous ethanol injection — HCC percutaneous ethanol injection
  Arms: percutaneous ethanol injection

SUMMARY:
Introduction: Liver transplantation(LT) is the gold-standard treatment for unresectable early-stage HCC within the Milan criteria. However, long waiting time can lead to dropout from LT candidacy. Local ablative procedures play a key role in the patient care enabling downsizing. Radiofrequency ablation(RFA) and percutaneous ethanol injection(PEI) are two valuable non-surgical neoadjuvant alternatives, but the most cost-effective treatment strategy remains controversial. Purpose: to assess whether RFA is cost-effective compared to PEI in adult patients with early-stage hepatocellular carcinoma within the Milan criteria. Methods: a pilot, single-center, randomized, open-label trial, with blinded end-point assessment, in which PEI was compared with RFA. Patients with early-stage hepatocellular carcinoma within the Milan criteria, listed for LT and indication for neoadjuvant treatment were eligible for enrollment. The primary outcome was the complete response rate according to mRECIST criteria at 60 days after the treatment. Secondary outcomes were the costs, rates and degrees of complications and the cost-effectiveness analysis of both techniques.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the fifth most common neoplasm worldwide, with more than 500,000 cases diagnosed annually. Its incidence has been increasing around the world, having doubled in the last 25 years in the United States and England. American statistics indicate that mortality from HCC is increasing compared to mortality from the vast majority of other types of cancer and it is estimated that mortality will double in the next two decades. In Brazil, an increasing trend in mortality was also observed for both sexes. The average mortality coefficient for the country was 3.59 deaths per 100 thousand inhabitants, with an annual linear increase of 0.020 (R2=0.588; p<0.001), being 4.20 deaths per 100 thousand men for males, with a linear increase of 0.044 (R2=0.81; p<0.001) per year and, for females, 2.98 per 100 thousand women, with an increase of 0.0194 (R2=0.35; p=0.008) per year.

The main etiological agents in the pathogenesis of HCC are chronic liver disease from chronic infection with hepatitis B (HBV) and hepatitis C (HCV) viruses and other causal factors of lower incidence such as alcohol abuse, metabolic/autoimmune disorders or environmental agents. Regarding HBV-mediated HCC, despite the availability of a vaccine against this virus, the World Health Organization estimates that, globally, 400 million people are chronically infected with HBV. There is no vaccine for HCV to date.

Proper diagnosis and treatment of HCC involves a multidisciplinary team comprised of oncologists, hepatologists, surgeons, pathologists, radiologists, and interventional radiologists. Currently, there are well-defined radiological criteria for the diagnosis of HCC, with biopsy being restricted to cases of diagnostic doubt. Multiphase cross-sectional imaging with contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI), or even contrast-enhanced ultrasound, allows for the non-invasive definitive diagnosis of HCC in patients considered to be at high risk. The Liver Imaging Reporting and Data System (universally known by its acronym LI-RADS - Liver Imaging Reporting and Data System), created in 2008 to address the need to improve the consistency and clarity of communication between radiologists and healthcare physicians. reference, has high specificity (above 85%) for patients at risk of HCC. Based on hyperenhancement in the arterial phase (HRFA), in addition to main criteria such as non-peripheral "washout", "capsule" with enhancement or growth above the threshold, suspicious nodules are categorized as probably HCC (LR-4) or definitely HCC , (LR-5).

Historically, radio and chemotherapy were not very effective in curing HCC and it was considered that surgical resection and liver transplantation were the only curative therapies in terms of disease-free survival for patients with HCC, but locoregional therapies such as ablation have become more effective in curing HCC. become potentially curative. Patients with preserved liver function or with lesions that require removal of a small non-tumorous liver mass are the best candidates for surgery. Unfortunately, only a minority of these patients can be candidates for surgery with definitive curative purposes, either due to the advanced stage of the disease at diagnosis, limitations in liver function, the presence of large, multiple tumors and/or located in an unfavorable location for safe resection.

The number of candidates for liver transplantation in relation to the limited supply of organs is still the main limiting factor for carrying out this procedure in our country. In Brazil, in May 2006, Ordinance No. 1160 modified the liver distribution criteria for transplants, implementing the severity criterion of the patient's clinical status, or model for end-stage liver disease (MELD - (MELD - mModel fFor Eend -sStage Liver Disease (MELD)), a scoring system that comprises a scale of values from 6 to 40, being considered a well-established method (AUC=0.78-0.87) as a predictor of three-month mortality in patients who are still on the waiting list for an organ. As an indicator of the severity of the recipient's end-stage biochemical dysfunction, the MELD score uses a logarithmic calculation that involves serum creatinine, bilirubin and International Normalized Ratio (INR), which evaluates the blood clotting tendency according to the formula: [0.957 x natural logarithm (Ln) (creatinine mg/dLl) + 0.378 x Ln (bilirubin mg/dlL) + 1.120 x Ln (INR) + 0.643] x 104.(6 ) Patients with HCC are classified as a special situation on the transplant list, with an initial MELD value of 20, as they are at a higher risk of death due to tumor progression, as well as the development of metastases or clinical decompensation, which can reach the maximum value of 29 after six months of inclusion on the list, if he has not been transplanted. Starting in 2016 in the United States and recently in Brazil, with the purpose of making the patient classification criteria increasingly more effective, it was proposed to adopt the serum sodium level in the MELD calculation (MELD-Na or MELD-sodium) , for the allocation of liver grafts. MELD-Na is calculated using the formula "MELD-Na=MELD + 1.32 x (137 - Na) - [0.033 x MELD*(137 - Na)]", considering the correction of the serum sodium value for the range of 125-137 mEq/lL and increasing the effectiveness in predicting mortality on the wait list. Another important factor considered when selecting patients with HCC for liver transplantation is the estimation of the risk of tumor recurrence in the post-surgical period. In current clinical practice in our country, this estimate is based on the size and number of tumor nodules and the presence of macroscopic vascular invasion, as defined in preoperative imaging studies. The rule proposed by the Milan group for patient selection, universally called the Milan Criteria (one nodule less than or equal to 5.0 cm or 2 to 3 nodules all less than or equal to 3.0 cm, and without macroscopic vascular invasion) has been shown to provide survival rates above 70% at 5 years with about a 10% probability of recurrence. These criteria have been validated by several groups and are widely used to select candidates in the United States and Europe. Despite its proven usefulness, however, it is well known that some patients with tumors exceeding these criteria are also potentially curable by liver transplantation. More recently, with the development of cell and molecular biology techniques, many molecular markers related to invasion, metastasis, recurrence and survival have been explored. In hepatocellular carcinomaHCC, DNA ploidy, proliferative activity of tumor cells, tumor suppressor and promoter genes, cell cycle controllers, proteinases that degrade the extracellular matrix, adhesion molecules, angiogenic factors and metabolic genes were considered biomarkers for the malignant phenotype of hepatocellular carcinoma, and are related to prognosis and therapeutic results.

The waiting time for liver transplantation in patients with HCC is a determining factor for a better prognosis, as disease progression can exclude them from the Milan Criteria and, consequently, from the transplant list. This progression rate varies from 7% to 11% in six months, and approaches 40% in one year. In these cases, it is understood that there is a loss of the criteria required to remain on the transplant list, with consequent exclusion of the patient from the waiting list, which is known as "drop-out" from the list. The waiting list time, which in other countries is around 6 months, in most regions of Brazil reaches more than a year and, sometimes, even with the special situation of patients with HCC on the list, the waiting time waiting time can exceed 2 years.

Over the past 30 years, several methods of chemical or thermal tumor destruction have been developed and clinically tested. Percutaneous ethanol injection (PEI) induces coagulative necrosis of the lesion as a result of cellular dehydration, protein denaturation and chemical occlusion of small tumor vessels. Later, thermal ablative therapies emerged and are classified as hyperthermic treatments (heating tissue to 60°-100°C) - including radiofrequency ablation (RFA). Most procedures are performed using a percutaneous approach guided by imaging methods, usually ultrasound and computed tomography.

It is notable that the principles of transplant benefit tend to prevail when the risk of cancer-related dropout and response to locoregional treatments are taken into account. Waitlisted candidates beyond accepted limits of transplantability are significantly more likely to die or be removed from the waitlist than less advanced candidates, but if prioritized and transplanted early show similar survival compared to hepatocellular carcinomaHCC less advanced.

There is consensus in the literature that neoadjuvant therapy finds its important role in reducing the risk of patients on the list within the Milan criteria, since if prioritized and maintained within the transplantability criteria they have similar survival regardless of whether or not they have hepatocellular carcinomaHCC. When analyzing the literature including patients not listed for transplantation, there are few randomized controlled studies that compare the best neoadjuvant therapy for hepatocellular carcinomaHCC.

A systematic review carried out in 2013 sought an answer to what would be the best treatment for patients with hepatocellular carcinomasHCC smaller than 3.0 cm, comparing radioblation (RFA) and percutaneous alcohol injection (PEI)RFA and PEI. They compiled evidence from 4 prospective randomized controlled studies, totaling 766 patients with follow-ups of at least 3 years. They concluded that RFA appears superior to PEI with regard to local tumor control and 3-year survival, but presents a greater number of complications and higher cost, being more feasible in patients with hepatocellular carcinomasHCC greater than 2.0 cm or with function hepatic Child-Pugh A.

Many patients in our country can certainly benefit from this modality, however, we do not yet have this treatment routinely available in Brazil given the potential high cost of the instrument, constant denials from supplementary paying sources and little availability in the public system. Hence the need for studies that aim to discuss conditions for the use of possible alternative technologies in our environment, such as percutaneous ethanol injection (PEI)PEI, which has a potential lower cost, but this cost has not yet been evaluated in our environment.

Patients on the liver transplant waiting list may benefit from percutaneous treatments involving RFA or PEI, but doubts remain as to whether PEI would have therapeutic disadvantages, fewer complications and a significantly lower cost compared to RFA.

The aim of this study is to compare the use of RFA with PEI in patients with hepatocellular carcinoma on the liver transplant waiting list, in relation to radiological response, complications, cost analysis and cost-effectiveness, as there is, to date, no sufficient evidence to uniformly support a better cost ratio and post-treatment tumor response considering the risk of complications, for RFA or PEI in HCCs between 2.0 and 3.0cm, especially in the national scenario.

It is also worth highlighting that there are no randomized controlled studies on the efficacy, cost-effectiveness and complications of RFA and PEI for patients with early-stage hepatocellular carcinomas on the liver transplant list in Latin America and very few randomized controlled studies published around the world.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of single or multiple HCC (up to three nodules), measuring between 2.0 and 3.0 cm according to the Barcelona Clinic Liver Cancer (tumor stage A) and Milan criteria.
* LI-RADS 4 or 5 nodule(s) evidenced on MRI for a maximum of 30 days, naïve to local treatment.
* Child-Pugh A and B patients on the liver transplant waiting list.

Exclusion Criteria:

* Presence of vascular invasion or extrahepatic dissemination;
* Refractory or intractable ascites;
* grade III/IV hepatic encephalopathy;
* Complete thrombosis of the main trunk of the portal vein;
* Total bilirubin >3mg/dlL;
* Coagulation disorder: INR>2 and/or platelets<20,000;
* Performance score (PST) according to the criteria of the Eastern Cooperative Oncology Group (ECOG) ECOG >2;
* Moderate or severe hydrothorax;
* Renal failure with creatinine clearance<30 mL/min/1.73 m²mlL/hr;
* Calculated MELD>30;
* Technical impediments to carrying out PEI or RFA procedures;
* Refusal to sign the Free and Informed Consent Term (TCLE);
* Patients who presented a greater risk with PEI or RFA procedures than the potential benefits of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
RFA versus PEI imaging response rate | 60 days
  To compare the objective response rate in magnetic resonance imaging performed approximately 60 days after radiofrequency ablation treatment or percutaneous alcohol injection as neoadjuvant therapy in patients with early-stage hepatocellular carcinomas (BCLC-A) on the waiting list for liver transplantation, according to mRECIST criteria.

SECONDARY OUTCOMES:
RFA versus PEI complication rate | 180 days
  Compare the rate of complications related to the methods
Compare the costs between RFA versus PEI | 180 days
  Compare the costs in US$ of radiofrequency ablation and percutaneous alcohol injection, from the day of the first intervention until the day of the last control MRI (180 days later).
late recurrenceof RFA versus PEI | 180 days
  Compare the late recurrences in MRIs between 120 and 180 days after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Mariotti, Principal Investigator — Hospital Israelita Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

REFERENCES:
- [Derived] Mariotti GC, Felga GEG, Garcia RG, Falsarella PM, Schmid BP, Malheiros DT, Baroni RH, Serpa Neto A. Cost-effectiveness of radiofrequency ablation versus percutaneous ethanol injection for early hepatocellular carcinoma in a resource-poor setting: a randomized trial. Einstein (Sao Paulo). 2024 Sep 30;22:eGS0683. doi: 10.31744/einstein_journal/2024GS0683. eCollection 2024. PMID 39356946